CLINICAL TRIAL: NCT05206487
Title: Hepatic Encephalopathy Prevention With Polydextrose After TIPS: Pilot Study
Brief Title: Hepatic Encephalopathy Prevention With Polydextrose After TIPS: Pilot Study (POEME)
Acronym: POEME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Société nationale française de gastro-entérologie (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/19/0493; 2020-A01217-32 (Other: ID-RCB)
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Hepatic Encephalopathy
Keywords: Hepatic Encephalopathy; TIPS; Microbiota; Polydextrose
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — polydextrose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polydextrose (Experimental): Patients will receive PDX 15 days prior and for a 6 month periods after TIPS.
  Interventions: Dietary Supplement: Polydextrose

INTERVENTIONS:
Dietary Supplement: Polydextrose — PDX will be started 2 weeks before TIPS and taken daily for a 6 month period after TIPS.

SUMMARY:
TIPS is a standard for the treatment of portal hypertension related complications. However, it remains at risk of HE after TIPS (around 40% the first year). Dysbiosis plays a key role in pathophysiology of HE.

Polydextrose (PDX) is consider as a prebiotic. Preliminary studies showed that PDX:

1. modified gut microbiota, enhancing "good bacteria"
2. improved gut permeability and immunity in 2 experimental models: infarction and colitis.

The aim of this study is to assess PDX efficacy to prevent HE during the first 6 months after TIPS in cirrhotic patients.

DETAILED DESCRIPTION:
TIPS is a standard for the treatment of portal hypertension related complications. However, it remains at risk of HE after TIPS (around 40% the first year). Dysbiosis plays a key role in pathophysiology of HE.

Polydextrose (PDX) is consider as a prebiotic. Preliminary studies showed that PDX:

1. modified gut microbiota, enhancing "good bacteria"
2. improved gut permeability and immunity in 2 experimental models: infarction and colitis.

Patients will receive PDX 15 days prior to and 6 months after TIPS. We will assess the cumulative incidence of HE 6 months after TIPS. Patients will be followed-up for 12 months after TIPS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age
* Affected (c) cirrhosis in which the establishment of a TIPS is scheduled within the month for: the treatment of ascites or a refractory hydrothorax or the prevention of the recurrence of a related digestive hemorrhage portal hypertension
* Having signed the consent to participate in the study
* Women of childbearing age on effective contraception
* Affiliated to a social security scheme

Exclusion Criteria:

* Contraindication for TIPS
* Digestive short circuit, chronic inflammatory bowel diseases
* Indications of TIPS in emergency or as part of the preparation for a surgical procedure,
* Liver transplant,
* Patient for whom the follow-up is considered impossible due to non-compliance with care or because the vital prognosis is estimated less than 6 months because of an incurable chronic pathology,
* Pregnant or lactating women,
* Those unable to receive enlightened information,
* Those participating in another interventional research including an exclusion period
* Persons placed under safeguard of justice, tutelage or curators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Hepatic encephalopathy incidence | 6 months
  The primary outcome is the cumulative incidence (%) of hepatic encephalopathy

SECONDARY OUTCOMES:
Number of patient with dose reduction | 6 months
  compliance will be evaluated by the number of patient with a dose reduction or who stop the product
Adverse events | 6 months
  safety will be evaluated by collection of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BUREAU, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bureau C, Metivier S, D'Amico M, Peron JM, Otal P, Pagan JC, Chabbert V, Chagneau-Derrode C, Procopet B, Rousseau H, Bosch J, Vinel JP. Serum bilirubin and platelet count: a simple predictive model for survival in patients with refractory ascites treated by TIPS. J Hepatol. 2011 May;54(5):901-7. doi: 10.1016/j.jhep.2010.08.025. Epub 2011 Feb 18. PMID 21145798
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines for the management of patients with decompensated cirrhosis. J Hepatol. 2018 Aug;69(2):406-460. doi: 10.1016/j.jhep.2018.03.024. Epub 2018 Apr 10. No abstract available. PMID 29653741
- [Background] Bureau C, Thabut D, Oberti F, Dharancy S, Carbonell N, Bouvier A, Mathurin P, Otal P, Cabarrou P, Peron JM, Vinel JP. Transjugular Intrahepatic Portosystemic Shunts With Covered Stents Increase Transplant-Free Survival of Patients With Cirrhosis and Recurrent Ascites. Gastroenterology. 2017 Jan;152(1):157-163. doi: 10.1053/j.gastro.2016.09.016. Epub 2016 Sep 20. PMID 27663604